CLINICAL TRIAL: NCT02511704
Title: Pharmacokinetics and Acute Effects of Multiple Dose of Nicotine Administered by Electronic Cigarette and Cigarette
Brief Title: Pharmacokinetics and Acute Effects of Multiple Dose of Nicotine: Electronic Cigarette and Cigarette
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Istituto Superiore di Sanità (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: IMIMFTCL/CIG-E/1
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2014-12

CONDITIONS: Nicotine Use Disorder
Keywords: Nicotine; Electronic cigarette; Cigarette
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic cigarette (Experimental): Multiple dose
  Nicotine 0.8 mg, administrated by electronic cigarette (10 puffs) + Nicotine 0.8 mg, administrated by electronic cigarette (10 puffs) separated by 60 minutes
  Interventions: Drug: Nicotine
- Cigarette (Active Comparator): Multiple dose
  Nicotine 0.8 mg, administrated by cigarette (10 puffs) + Nicotine 0.8 mg, administrated by cigarette (10 puffs) separated by 60 minutes
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Multiple dose nicotine
  Other Names: Nhoss®
  Arms: Electronic cigarette
Drug: Nicotine — Multiple dose nicotine
  Other Names: Marlboro®
  Arms: Cigarette

SUMMARY:
The purposes of this study are 1) to determine the pharmacokinetics of nicotine after multiple dose administration by electronic cigarette and 2) to compare the acute effects of multiple dose of nicotine administrated by electronic cigarette compared with those obteined by cigarette.

DETAILED DESCRIPTION:
Electronic cigarettes (e-cigarettes) are battery-operated devices that deliver nicotine via inhaled vapour or "vaping". At present, e-cigarettes are becoming increasingly popular among smokers worldwide. However, knowledge about e-cigarette nicotine pharmacology remains limited.

The aims of this study are 1) to determine the pharmacokinetics of nicotine after multiple dose administration by electronic cigarette and 2) to compare the acute effects of multiple dose of nicotine administrated by electronic cigarette compared with those obteined by cigarette.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting the study procedures and signing the informed consent.
* Male adults volunteers (18-45 years old).
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* Present use of nicotine without serious adverse reactions.
* Smokers ≥ 3 cigarettes/day.

Exclusion Criteria:

* Having suffered any cardiovascular and/or respiratory disease in the three months prior to the study start.
* History of drug dependence (except for nicotine dependence).
* Daily consumption >4 standard units of ethanol.
* Regular use of any drug in the month prior to the study sessions. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* Blood donation 12 weeks before or participation in other clinical trials with drugs in the previous 12 weeks.
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Use of any drug or substance inhibitor of cytochrome P-450-1A6 (CYP1A6) (p.e. raloxifene, coumarins, etc)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-24h) | From baseline (pre-dose, 0h) to 5, 15, 30, 45, 55, 65, 75, 90, 105, 120 and 24h post-dose
  Calculation of AUC of the concentrations of nicotine and its metabolites in blood

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-24h) | From baseline (pre-dose, 0h) to 55, 120 min, 6, 12 and 24h
  Calculation of AUC of the concentrations of nicotine and its metabolites in urine
Area Under the Concentration-Time Curve (AUC 0-24h) | From baseline (pre-dose, 0h) to 15, 30, 45, 55, 65, 75, 90, 105, 120 min, 6, 12 and 24h
  Calculation of AUC of the concentrations of nicotine and its metabolites in oral fluid
Number of Participants with Serious and Non-Serious Adverse Events | 2 days after each substance administration
  Collection of adverse effects spontaneously reported by the participants and/or observed by the investigators
Elimination half-life | From baseline to 24h post-dose
  Calculation of elimination hal-life from concentrations of nicotine and its metabolites in plasma-blood, urine and oral fluid.
Changes in blood pressure | From pre-dose (baseline) to 120 min post-dose
  Measure of blood pressure (systolic and diastolic blood pressure)
Changes in heart rate | From pre-dose (baseline) to 120 min post-dose
  Measure of heart rate (pulse)
Changes in expired carbon monoxide (CO) aire | From pre-dose (baseline) to 120 min post-dose
  Measure of expired CO aire using a BreathCO monitor
Changes in pupil diameter | From pre-dose (baseline) to 120 min post-dose
  Measure of pupil diameter using a Haab pupil gauge
Changes in oral temperature | From pre-dose (baseline) to 120 min post-dose
  Measure of temperature in mouth using automatic thermometer
Changes in subjective effects | From pre-dose (baseline) to 120 min post-dose
  Subjective effects will be measured using rate scales (visual analogue scales) including measures of good effects and other feelings induced by nicotine
Changes in nicotine abstinence symptoms | From pre-dose (baseline) to 120 min post-dose
  Nicotine abstinence symptoms will be measured using rate scales (visual analogue scales) including items sensitive to nicotine effects

CONTACTS AND LOCATIONS:
Overall Officials: Magi Farre, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Institut Hospital del Mar d'Investigacions Mèdiques-IMIM. Parc de Salut Mar., Barcelona, Barcelona, Spain